CLINICAL TRIAL: NCT05767437
Title: The Effects of Reaching Task Following Selective Trunk Stability Exercise in Chronic Stroke Survivors
Brief Title: The Effects of Reaching Task Following Selective Trunk Stability Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ulsan National Institute of Science and Technology (Unknown)
Responsible Party: Principal Investigator, José Casaña Granell, Professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ADIM exercise
Record Dates: First submitted 2022-12-23; First posted 2023-03-14 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Stroke; Hemiplegia, Spastic
Keywords: Reaching task; Abdominal drawing-in maneuver; ADIM; Chronic stroke
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: One group is the abdominal drawing-in maneuver exercise, afterward conventional physiotherapy in Participants With stroke survivors. On the contrary, Another group is conventional physiotherapy afterward the abdominal drawing-in maneuver exercise.
Who Masked: Participant, Investigator
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal drawing-in maneuver exercise, afterward Sham therapy(conventional physiotherapy) (Experimental): Participants first received Abdominal drawing-in maneuver exercise 2 times a week for 4 weeks. Each session is 40 minutes for additional 10 min with conventional therapy. Afterward a washout period of one month, they then received sham therapy (conventional therapy_release pain or upper limb mobilization) 2 times a week for 4 weeks. Each session is 40 minutes.
  Interventions: Behavioral: Abdominal drawing-in maneuver exercise; Behavioral: sham
- Sham therapy(conventional physiotherapy), afterward Abdominal drawing-in maneuver exercise (Experimental): Participants first received sham therapy(release pain or upper limb mobilization)2 times a week for 4 weeks. Each session is 40 minutes. Afterward a washout period of one month, they then received Abdominal drawing-in maneuver exercise 2 times a week for 4 weeks. Each session is 40 minutes for additional 10 min with conventional therapy
  Interventions: Behavioral: Abdominal drawing-in maneuver exercise; Behavioral: sham

INTERVENTIONS:
Behavioral: Abdominal drawing-in maneuver exercise — From the supine position to the hook-lying position (hip joint at 40 degrees and the knee joint at 80 degrees) and pull the navel deeply to the lumbar region through the Stabilizer™ Pressure Biofeedback that stabilize transversus abdominis muscle. At this time, subjects are controlled to maintain contraction while keep breathing lightly, to contract slowly, also to not move the pelvis and chest while exercising
  Other Names: Stabilizer pressure biofeedback
Behavioral: sham — Release pain or upper limb mobilization
  Other Names: Conventional therapy

SUMMARY:
This study is performed in a controlled randomized, two-period crossover design to test the efficacy of Abdominal drawing-in maneuver (ADIM) exercise compared to conventional physiotherapy in chronic stroke survivors.

DETAILED DESCRIPTION:
All participants provided written informed consent and are assigned to Group A or Group B. The inclusion criteria are Exclusion criteria are

Abdominal drawing-in maneuver exercise is following as:

It's for strengthening the Transversus Abdominis muscle(TrA). The simple device, that observes the pressure changes by the gauge. Subjects receive intervention 2 times a week for 4 weeks. Each session is 40 minutes. From the supine position to the hook-lying position (hip joint at 40 degrees and the knee joint at 80 degrees) and pull the navel deeply to the lumbar region through the Stabilizer™ Pressure Biofeedback that stabilizes transversus abdominis muscle. At this time, subjects are controlled to maintain contraction while keep breathing lightly, to contract slowly, also to not move the pelvis and chest while exercising The device assists in body control movements of the spine and abdominal muscle.

Conventional physiotherapy is following as:

Release pain, limb stretching, mobilization of joint and pelvic movement. Subjects receive 2 times a week for 4 weeks. Each session is 40 minutes. Group A received Abdominal drawing-in maneuver exercise for 4 weeks on period 1. Afterward washout period in a month, follow period 2 of conventional physiotherapy.

On the other side, Group B receives first conventional physiotherapy on period 1. Afterward washout period in a month, follow period 2 of Abdominal drawing-in maneuver exercise.

ELIGIBILITY:
Inclusion Criteria:

* The subject consisted of the physician's confirmation of chronic hemiplegia
* onset ≥ 6 months
* Mini-mental state examination≥25
* Biceps ≤2, Triceps≤2
* Ability to Sit on a chair alone
* FMA UE score ≥ 21points, FMA UE≤ 60 points

Exclusion Criteria:

* Biceps>2, Triceps>2
* Flaccid
* Neglect syndrome
* Have neurological disease and orthopedic disease
* Lack of coordination

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jóse Casaña Granell, PhD, Principal Investigator — University of Valencia; Joaquin Calatayud Villalba, PhD, Principal Investigator — University of Valencia; Sang Hoon Kang, PhD, Principal Investigator — Ulsan National Institute of Science&Technology
Locations (1):
- Ulsan National Institute of Science and Technology, Ulsan, Ulju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messier S, Bourbonnais D, Desrosiers J, Roy Y. Dynamic analysis of trunk flexion after stroke. Arch Phys Med Rehabil. 2004 Oct;85(10):1619-24. doi: 10.1016/j.apmr.2003.12.043. PMID 15468021
- [Background] Cirstea MC, Levin MF. Compensatory strategies for reaching in stroke. Brain. 2000 May;123 ( Pt 5):940-53. doi: 10.1093/brain/123.5.940. PMID 10775539
- [Background] Velozo CA, Woodbury ML. Translating measurement findings into rehabilitation practice: an example using Fugl-Meyer Assessment-Upper Extremity with patients following stroke. J Rehabil Res Dev. 2011;48(10):1211-22. doi: 10.1682/jrrd.2010.10.0203. PMID 22234665
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] Lee PY, Huang JC, Tseng HY, Yang YC, Lin SI. Effects of Trunk Exercise on Unstable Surfaces in Persons with Stroke: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Dec 7;17(23):9135. doi: 10.3390/ijerph17239135. PMID 33297451
- [Background] Kelli A, Kellis E, Galanis N, Dafkou K, Sahinis C, Ellinoudis A. Transversus Abdominis Thickness at Rest and Exercise in Individuals with Poststroke Hemiparesis. Sports (Basel). 2020 Jun 12;8(6):86. doi: 10.3390/sports8060086. PMID 32545550
- [Result] Haruyama K, Kawakami M, Otsuka T. Effect of Core Stability Training on Trunk Function, Standing Balance, and Mobility in Stroke Patients. Neurorehabil Neural Repair. 2017 Mar;31(3):240-249. doi: 10.1177/1545968316675431. Epub 2016 Nov 9. PMID 27821673
- [Result] Wu CY, Liing RJ, Chen HC, Chen CL, Lin KC. Arm and trunk movement kinematics during seated reaching within and beyond arm's length in people with stroke: a validity study. Phys Ther. 2014 Jun;94(6):845-56. doi: 10.2522/ptj.20130101. Epub 2014 Jan 30. PMID 24481598

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants dropped out during the washout period, leading to a smaller sample size and uneven group distribution in period 2.
Period: Overall Study
Arm/Group | Abdominal drawing-in Maneuver Exercise, Afterward Sham Therapy(Conventional Physiotherapy) | Sham Therapy(Conventional Physiotherapy), Afterward Abdominal drawing-in Maneuver Exercise
Started | 10 | 10
Completed | 10 | 6
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: Upper limb impairment was evaluated using the Fugl-Meyer Assessment, which categorized participants based on the severity of impairment. To assess spasticity in the elbow flexor and extensor muscles, the Modified Ashworth Scale (MAS) was used. Postural control of the upper limb was assessed using the Postural Assessment Scale for Stroke (PASS). The Trunk Impairment Scale (TIS) was also employed to evaluate static and dynamic sitting balance and coordination. Range of motion (ROM) was assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal drawing-in Maneuver Exercise, Afterward Sham Therapy(Conventional Physiotherapy) | Sham Therapy(Conventional Physiotherapy), Afterward Abdominal drawing-in Maneuver Exercise | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.20 (10.05) | 60.83 (10.55) | 66.69 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: scores on subscale] — Measure Description: Inclusion criteria: FMA upper extremity score < 60 points (In sitting position, the sum of each subtotal score is 66 (maximum) and the minimum is 0. Subscales were summed to compute a total score. Cutoff scores defined 0~20: severe, 21 ~ 50: moderate, 51~66: mild
  1) Reflex activity_max 4 score, 2) Volitional movement within synergies_ max 18, 3) Volitional movement mixing synergies_ max 6, 4) Volitional movement with little or no synergy_ max 6, 5) Normal reflex activity_max 2, 6) Wrist movement_ max 10, 7) Hand movement with grasp_ max 14, 8) coordination/speed_max 6.
  scores on subscale | 36.90 (15.47) | 40.00 (11.95) | 38.06 (13.91)
Onset [Mean (Standard Deviation); unit: Months] | 157.70 (119.59) | 142.00 (78.16) | 151.81 (103.34)
Height [Mean (Standard Deviation); unit: centimeter] | 160.00 (4.90) | 164.58 (7.93) | 161.72 (6.37)
Side of paralysis [Count of Participants; unit: Participants]
  Left | 5 | 2 | 7
  Right | 5 | 4 | 9
Postural Assessment Scale for Stroke [Mean (Standard Deviation); unit: units on a scale] — The Postural Assessment Scale for Stroke (PASS) evaluates postural control in stroke patients, with scores ranging from 0-36 points, where higher scores indicate better functional recovery.
  1) Sitting without support 2,3) Standing with(without) support 4,5) Standing on (non)paretic leg 6) Supine to affected side lateral 7) Supine to non-affected side lateral 8) Supine to sitting up on the edge of the table 9) Sitting on the edge of the table to supine 10) Sitting to standing up 11) Standing up to sitting down 12) Standing, picking up a pencil from the floor
  units on a scale | 33.30 (2.36) | 30.33 (4.76) | 32.19 (3.62)
Trunk Impairment Scale for stroke [Mean (Standard Deviation); unit: units on a scale] — The Trunk Impairment Scale (TIS) for stroke has a total score of 23 points, with higher scores indicating better trunk control ability. TIS components:
  Static sitting balance - 7 points Dynamic sitting balance - 10 points Coordination - 6 points 23 points = Optimal trunk control ability (normal performance of all items) 0 points = Minimal trunk control ability (unable to perform)
  1. Static sitting balance
  2. Dynamic sitting balance
  3. Co-ordination
  units on a scale | 14.40 (3.98) | 14.50 (5.32) | 14.44 (4.35)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of a Particular Intervention During the Entire Course of the study_Trunk Dislocation
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10%.
  Participants who received that particular intervention during the entire course of the study. Effect of Abdominal Drawing-In Maneuver (AIDM) exercise and Shan therapy. Dislocation distance in millimeters(mm) for reaching phase
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: Patients were randomly assigned to either Group A or Group B.
Measure: Mean (Standard Deviation); unit: Millimeter
Groups:
- Abdominal drawing-in Maneuver Exercise: Participants first received Abdominal drawing-in maneuver exercise 2 times a week for 4 weeks. Each session is 40 minutes for additional 10 min with conventional therapy. Afterward a washout period of one month, they then received sham therapy (conventional therapy_release pain or upper limb mobilization) 2 times a week for 4 weeks. Each session is 40 minutes.
  Abdominal drawing-in maneuver exercise: From the supine position to the hook-lying position (hip joint at 40 degrees and the knee joint at 80 degrees) and pull the navel deeply to the lumbar region through the Stabilizer™ Pressure Biofeedback that stabilize transversus abdominis muscle. At this time, subjects are controlled to maintain contraction while keep breathing lightly, to contract slowly, also to not move the pelvis and chest while exercising
  sham: Release pain or upper limb mobilization
- Sham Therapy(Conventional Physiotherapy): Participants first received sham therapy(release pain or upper limb mobilization)2 times a week for 4 weeks. Each session is 40 minutes. Afterward a washout period of one month, they then received Abdominal drawing-in maneuver exercise 2 times a week for 4 weeks. Each session is 40 minutes for additional 10 min with conventional therapy
  Abdominal drawing-in maneuver exercise: From the supine position to the hook-lying position (hip joint at 40 degrees and the knee joint at 80 degrees) and pull the navel deeply to the lumbar region through the Stabilizer™ Pressure Biofeedback that stabilize transversus abdominis muscle. At this time, subjects are controlled to maintain contraction while keep breathing lightly, to contract slowly, also to not move the pelvis and chest while exercising
  sham: Release pain or upper limb mobilization
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
Millimeter | 304.97 (83.22) | 303.34 (45.74)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — effect size of 0.02, α < 0.05, power = 0.02; p = 0.98, Mixed Models Analysis; Mean Difference (Net) = 1.63, 95% CI 2-sided [-55.79 to 59.05]

2. Primary Outcome: The Effect of a Particular Intervention During the Entire Course of the Study_movement Unit
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10%.
  It was defined by velocity peaks exceeding 20mm/s, with a minimum 150 ms interval.
  Participants who received that particular intervention during the entire course of the study.
  Number of movement units for reaching phase
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: Number of movements
Groups:
- Sham Therapy(Conventional Therapy): Participants first received sham therapy(release pain or upper limb mobilization)2 times a week for 4 weeks. Each session is 40 minutes. Afterward a washout period of one month, they then received Abdominal drawing-in maneuver exercise 2 times a week for 4 weeks. Each session is 40 minutes for additional 10 min with conventional therapy
  Abdominal drawing-in maneuver exercise: From the supine position to the hook-lying position (hip joint at 40 degrees and the knee joint at 80 degrees) and pull the navel deeply to the lumbar region through the Stabilizer™ Pressure Biofeedback that stabilize transversus abdominis muscle. At this time, subjects are controlled to maintain contraction while keep breathing lightly, to contract slowly, also to not move the pelvis and chest while exercising
  sham: Release pain or upper limb mobilization
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Therapy)
Number analyzed (Participants) | 16 | 16
Number of movements | 4.30 (1.60) | 4.30 (1.39)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Therapy); Test type: Equivalence — an effect size of 0.00, α < 0.05, power = 0.00; p = 0.99, Mixed Models Analysis; Mean Difference (Net) = 0.00, 95% CI 2-sided [-1.25 to 1.24]

3. Primary Outcome: The Effect of a Particular Intervention During the Entire Course of the Study_Elbow Angle
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10% Elbow angle in degree for reaching phase Participants who received that particular intervention during the entire course of the study.
  -elbow angle: joining vector of acromion to lateral epicondyle and vector of lateral epicondyle and medial styloid process.
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: degree on angle
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
degree on angle | 127.43 (25.23) | 134.13 (13.89)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — an effect size of 0.56 , α < 0.05, power = 32.5; p = 0.68, Mixed Models Analysis; Mean Difference (Net) = 6.71, 95% CI 2-sided [-24.12 to 10.71]

4. Secondary Outcome: The Effect of a Particular Intervention During the Entire Course of the Study_Total Time
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10%.
  Participants who received that particular intervention during the entire course of the study.
  Duration of time in second(s) for reaching phase
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: Second on time
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
Second on time | 3.25 (0.78) | 3.06 (0.88)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); an effect size of 0.24, α < 0.05, power = 24.5; Test type: Equivalence — Analysis population description: patients were randomly assigned to either Group A or Group B; p = 0.56, Mixed Models Analysis; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.48 to 0.87]

5. Secondary Outcome: The Effect of a Particular Intervention During the Entire Course of the Study_Hand Velocity
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10%.
  Participants who received that particular intervention during the entire course of the study.
  We analyzed peak hand velocity (mm/s) as velocity per unit time
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: Millimeter per second on time
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
Millimeter per second on time | 684.13 (339.62) | 934.48 (560.00)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — an effect size of 0.56, α < 0.05, power = 57.9; p = 0.42, Mixed Models Analysis — Interaction of Assessment and Group; Mean Difference (Net) = -250.35, 95% CI 2-sided [-614.88 to 114.18]

6. Secondary Outcome: The Effect of a Particular Intervention During the Entire Course of the Study_Elbow Angular Velocity
Description: We defined hand movement onset as the time when tangential velocity exceeded 10% of peak velocity and movement offset as when it fell below 10%.
  Participants who received that particular intervention during the entire course of the study.
  Peak angular velocity (rad/s) for the elbow were assessed during extension.
Time Frame: Baseline, two period(each 4weeks), wash out(4weeks)
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: Degree per second on time
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
Degree per second on time | 54.23 (50.83) | 41.98 (27.79)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — an effect size of 0.29, α < 0.05, power = 88.9; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = 12.25, 95% CI 2-sided [-18.67 to 43.17]

7. Other Pre Specified Outcome: Modified Ashworth Scale(MAS)_Stiffness of Chronic Stroke
Description: Scoring for Biceps and Triceps
  * MAS 0: No increase in tone
  * MAS 1: slight increase in tone giving a catch when slight increase in muscle t-tone, manifested by the limb was moved in flexion or extension.
  * MAS 1+: slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM )
  * MAS 2: more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  * MAS 3: considerable increase in tone, passive movement difficult
  * MAS 4: limb rigid in flexion or extension (MAS grade of 1 is equivalent to 1, whereas a MAS grade of 1+ includes grade of 2, 2->3, 3->4 in our study)
Time Frame: Baseline
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
Score on a scale | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — an effect size of 0.18, α < 0.05, power =6.5; p = 0.67, Wilcoxon (Mann-Whitney) — MAS of Biceps; mean rank (Z) = 0.18, 95% CI 2-sided [-0.61 to 0.96]

8. Other Pre Specified Outcome: Fugl Meyer Assessment(FMA)_Health Status Chronic Stroke
Description: Upper extremity(UE) Commonly used FMA-UE cutoff scores defined each category: 0 to 20 severe, 21 to 50 moderate, and 51 to 66 mild.
  * Shoulder, Elbow and Forearm
    1. Reflex activity
    2. Volitional movement within synergies
    3. Volitional movement mixing synergies
    4. Volitional movement with little or no synergy
    5. Normal reflex activity
  * Wrist
  * Hand
  * Coordination/Speed Total score is 66 points
Time Frame: Baseline
Population: Analysis population description: patients were randomly assigned to either Group A or Group B
Measure: Mean (Standard Deviation); unit: score on a subscale
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
Number analyzed (Participants) | 16 | 16
score on a subscale | 42.73 (18.94) | 49.36 (14.23)
Statistical Analysis 1: Comparison: Abdominal drawing-in Maneuver Exercise vs Sham Therapy(Conventional Physiotherapy); Test type: Equivalence — an effect size of 0.39, α < 0.05, power = 16.2; p = 0.38, t-test, 2 sided; Mean Difference (Net) = -6.63, 95% CI 2-sided [-19.38 to 6.12]

ADVERSE EVENTS:
Time Frame: 4 weeks after baseline measurement and after 4 weeks after period 2
Description: Participants were monitored during exercise sessions for potential adverse events. Due to the nature of the basic abdominal exercises with conventional physiotherapy implemented in this study, no adverse events (including all-cause mortality, serious adverse events, or other adverse events) were observed or reported. The low-risk nature of the basic abdominal exercises with conventional physiotherapy contributed to this outcome.
  Adverse events were monitored/assessed, but none were observed
Arm/Group | Abdominal drawing-in Maneuver Exercise | Sham Therapy(Conventional Physiotherapy)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal drawing-in Maneuver Exercise (N=16) | Sham Therapy(Conventional Physiotherapy) (N=16)
Other (Not including Serious) Adverse Events (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal drawing-in Maneuver Exercise (N=16) | Sham Therapy(Conventional Physiotherapy) (N=16)
Temporal discomfort (Investigations) | 0 (0) | 0 (0) — 1. Localized pruritus 2. abdominal discomfort

LIMITATIONS AND CAVEATS:
we must acknowledge a limitation in our study related to the influence of a carryover effect and period effect. This phenomenon may be partially explained within the context of persistence of treatment and learned behavior. Secondly, our study employed a crossover design, spanning a three-month duration. Despite random allocation, four participants dropped out during the washout period, leading to a smaller sample size and uneven group distribution in period 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT05767437/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05767437/SAP_001.pdf